CLINICAL TRIAL: NCT01937611
Title: Comparison of Dexmedetomidine and Midazolam as Intramuscular Premedication for Suspension Laryngoscopy
Brief Title: Intramuscular Dexmedetomidine as Premedication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, Professor, Deputy Director, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20121A021007
Record Dates: First submitted 2013-09-01; First posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Laryngoscopy; Preanesthetic Medication
Keywords: dexmedetomidine; intramuscular premedication; bradycardiac
MeSH Terms: interventions — Dexmedetomidine; Therapeutics; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): dexmedetomidine 1μg•kg-1
  Interventions: Drug: Dexmedetomidine
- midazolam (Active Comparator): midazolam 0.03 mg•kg-1
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine
  Other Names: Treatment
  Arms: Dexmedetomidine
Drug: Midazolam — Midazolam
  Other Names: control
  Arms: midazolam

SUMMARY:
Many studies have been conducted for the feasibility of using dexmedetomidine as premedication. However, bradycardia and hypotension frequently occurred following the premedication with dexmedetomidine, either via intramuscular or intravenous route. This is particularly true when using a high dose of dexmedetomidine: a intramuscular dose over 2 μg•kg-1 or a intravenous dose over 1 μg•kg-1 can elicit marked decreases in heart rate and mean arterial blood pressure. Subsequent studies using high-dose dexmedetomidine further revealed the potential impact of its detrimental haemodynamic profile on clinical outcomes. Most studies using high-dose dexmedetomidine were predominantly adopted with the dose-finding study performed by Aho and colleague, whom reported that 2.5 μg•kg-1 dose of intramuscular dexmedetomidine was comparably sedative and anxiolytic to 0.08 mg•kg-1 midazolam. However, few investigations have addressed the clinical effects of low-dose dexmedetomidine as premedication. Considering modern anaesthesia has advanced a long way towards eliminating the routine need for a deep preoperative sedation. It has, therefore, become desirable to asses dexmedetomidine as an effective premedication using a moderate sedative dose to minimize its undesired hemodynamic effects. We set a prospective study to compare the sedative, haemodynamic, adjuvant anaesthetic effects and patient's satisfaction of low-dose dexmedetomidine (1μg•kg-1) with midazolam (0.03 mg•kg-1), the most commonly used premedication, used as an intramuscular injective administration in patients undergoing suspension laryngoscopic surgery under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-55 years old, American Society of Anaesthesiologists physical status I, scheduled for elective suspension laryngoscopic surgery of benign vocal fold lesions.

Exclusion Criteria:

* Patients with neurological deficits
* Pregnancy
* Imprisonment
* Morbid obesity (body mass index ≥ 30 kg•m-2)
* Preoperative heart rate <45 beats•min-1
* Second or third degree atrioventricular block
* Antihypertensive medication with α-methyldopa, clonidine or other α2-adrenergic agonist

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Perioperative heart rate response | Participants will be monitored for the duration of anesthesia and recovery, an expected average of 2 hours.

SECONDARY OUTCOMES:
Sedation | Participants will be monitored for the duration of anesthesia and recovery, an expected average of 2 hours.
Adjuvant anesthesia effect | Participants will be monitored for the duration of anesthesia, an expected average of half an hour.
  Target-controlled infusion concentrations of propofol and remifentanyl at intubation, start and completion of surgery.
Patient's over-all satisfaction | On leaving the post-care unite, an expected average of 2 min.
  On discharge from recovery patients were asked to rate their satisfaction with the anaesthesia and the surgery that they had received as; highly satisfactory, acceptable, or unacceptable.

OTHER OUTCOMES:
Mean arterial blood pressure | Participants will be monitored for the duration of anesthesia and recovery, an expected average of 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PhD., Principal Investigator — Affiliated First People's Hospital of Guangzhou, Guangzhou Medical University
Locations (1):
- Affiliated First People's Hospital of Guangzhou, Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Jayaraman L, Sinha A, Punhani D. A comparative study to evaluate the effect of intranasal dexmedetomidine versus oral alprazolam as a premedication agent in morbidly obese patients undergoing bariatric surgery. J Anaesthesiol Clin Pharmacol. 2013 Apr;29(2):179-82. doi: 10.4103/0970-9185.111680. PMID 23878437
- [Result] Gupta K, Jain M, Gupta PK, Rastogi B, Saxena SK, Manngo A. Dexmedetomidine premedication for fiberoptic intubation in patients of temporomandibular joint ankylosis: A randomized clinical trial. Saudi J Anaesth. 2012 Jul;6(3):219-23. doi: 10.4103/1658-354X.101211. PMID 23162393
- [Result] Mowafi HA, Aldossary N, Ismail SA, Alqahtani J. Effect of dexmedetomidine premedication on the intraocular pressure changes after succinylcholine and intubation. Br J Anaesth. 2008 Apr;100(4):485-9. doi: 10.1093/bja/aen020. Epub 2008 Feb 19. PMID 18285392
- [Result] Peden CJ, Cloote AH, Stratford N, Prys-Roberts C. The effect of intravenous dexmedetomidine premedication on the dose requirement of propofol to induce loss of consciousness in patients receiving alfentanil. Anaesthesia. 2001 May;56(5):408-13. doi: 10.1046/j.1365-2044.2001.01553.x. PMID 11350323
- [Result] Taittonen MT, Kirvela OA, Aantaa R, Kanto JH. Effect of clonidine and dexmedetomidine premedication on perioperative oxygen consumption and haemodynamic state. Br J Anaesth. 1997 Apr;78(4):400-6. doi: 10.1093/bja/78.4.400. PMID 9135361
- [Result] Erkola O, Korttila K, Aho M, Haasio J, Aantaa R, Kallio A. Comparison of intramuscular dexmedetomidine and midazolam premedication for elective abdominal hysterectomy. Anesth Analg. 1994 Oct;79(4):646-53. doi: 10.1213/00000539-199410000-00006. PMID 7943770
- [Result] Virkkila M, Ali-Melkkila T, Kanto J, Turunen J, Scheinin H. Dexmedetomidine as intramuscular premedication for day-case cataract surgery. A comparative study of dexmedetomidine, midazolam and placebo. Anaesthesia. 1994 Oct;49(10):853-8. doi: 10.1111/j.1365-2044.1994.tb04257.x. PMID 7802178
- [Derived] Sun Y, Liu C, Zhang Y, Luo B, She S, Xu L, Ruan X. Low-dose intramuscular dexmedetomidine as premedication: a randomized controlled trial. Med Sci Monit. 2014 Dec 18;20:2714-9. doi: 10.12659/MSM.891051. PMID 25529851